CLINICAL TRIAL: NCT04182854
Title: Use of Diuretics in Maintenance Hemodialysis Patients With Residual Renal Function Undergoing Bioimpedance-guided Fluid Management
Brief Title: Use of Diuretics in Maintenance Hemodialysis Patients Undergoing Bioimpedance-guided Fluid Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Dongliang Zhang, MD, professor, Peking University International Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YN2017QN15
Record Dates: First submitted 2019-11-22; First posted 2019-12-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Diuretic Abuse
Keywords: furosemide; hydrochlorothiazide; residual renal function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- diuretics (Experimental)
  Interventions: Drug: Furosemid hydrochlorothiazide

INTERVENTIONS:
Drug: Furosemid hydrochlorothiazide — furosemide 100mg for one month;furosemide 200mg for one month;furosemide 100mg and hydrochlorothiazide 25mg for one month;

SUMMARY:
Background.The objective of the present study is to verify whether using diuretics will improve either blood pressure or fluid overload in maintenance hemodialysis patients with residual diuresis kidney function.

DETAILED DESCRIPTION:
Methods.46 maintenance hemodialysis patients will be given three stages of diuretic intervention: 100mg furosemide every day for 1 month, 200mg furosemide every day for 1 month, and 100mg furosemide combined with 25mg hydrochlorothiazide every day for 1 month. The 24-hour urine volume, 24-hour urine sodium, 24-hour urine potassium, blood pressure, OH(overhydration) and dry weight will be collected. OH will be measured by bioelectrical impedance.

ELIGIBILITY:
Inclusion Criteria:

* maintenance hemodialysis patient
* unrine volume more than 100ml.

Exclusion Criteria:

* myocardial infarction;
* unrine volume less than 100ml.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
urine volume increasing after diuretic use in maintenance hemodialysis patients with residual renal function | up to 16 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University internation Hospital, Beijing, Beijing Municipality, China